CLINICAL TRIAL: NCT05816395
Title: A Randomized, Placebo Controlled, Investigator and Participant-blinded Study Investigating Safety, Tolerability, and Efficacy of RHH646 in Participants With Knee Osteoarthritis
Brief Title: Safety and Efficacy of RHH646 for Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRHH646A12201; 2022-502821-16-00 (Other: CTIS)
Record Dates: First submitted 2023-01-31; First posted 2023-04-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Knee
Keywords: Tibiofemoral OA; K&L grade 2 to 3 OA in the target knee; Oral RHH646 treatment
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RHH646 (Experimental): RHH646
  Interventions: Drug: RHH646
- Placebo (Placebo Comparator): RHH646 placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RHH646 — RHH646 capsule for oral use
  Arms: RHH646
Drug: Placebo — RHH646 placebo capsule for oral use
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the articular cartilage-regenerating capacity of RHH646 in the knee as well as to assess safety and tolerability in participants with knee osteoarthritis. The treatment duration will be up to 52 weeks. The total study duration for an individual participant will be up to 62 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≥35 and ≤75 years old, at time of screening
* Participants must weigh at least 50 kg to participate in the study and must have a body mass index (BMI) ≤35 kg/m2. BMI = Body weight (kg) / [Height (m)]2
* Diagnosis of tibiofemoral OA in at least one knee by standard American College of Rheumatology clinical and radiographic criteria (Altman et al 1986) at screening
* K&L grade 2 to 3 OA in the target knee evaluated with X-Ray by the Central Reader at screening
* Predominantly medial tibiofemoral compartment involvement defined as medial Joint Space Narrowing (medJSN) 1-2 (Altman et al 1995; Altman, Gold 2007) and medJSN > lateral Joint Space Narrowing (latJSN) in the target knee evaluated with X-Ray by the Central Reader at screening
* Symptomatic disease, defined as having pain in the target knee at least 3 days per week during the last 3 months from screening that is relieved by analgesic therapy (e.g. acetaminophen or non-steroidal anti-inflammatory drugs), according to the investigator's evaluation and judgment of the patient's history

Exclusion Criteria:

* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception. In EEA countries, women of child-bearing potential will be excluded from participation in this trial, irrespective of the use of highly effective methods of contraception.
* Arthroscopy of the target knee within the 6 months prior to screening or planned arthroscopy during the study
* Previous surgical treatment of the target knee using mosaicplasty, microfracture, meniscectomy >50% or osteotomy; planned surgery for either knee during the study
* Unstable target knee joint (including, but not limited to, post-traumatic or congenital laxity) or insufficiently reconstructed ligaments based on medical history and/or physical examination by the investigator
* Participant has severe malalignment (valgus or varus deformity) in the target knee >7.5° based on X-ray evaluation by the Central Reader at screening.
* K&L grade 4 OA in either knee
* Presence of severe hip OA that either (i) alters lower limb function to a degree that increases or abnormally changes the mechanical forces in the knee while walking, according to investigator's evaluation or (ii) currently requires or is likely to require specific medical or surgical management during the study period
* Other pathologies affecting the knee, including subchondral insufficiency fractures, bone fracture (acute or subacute within the 6 months prior to screening) or bone bruise, osteonecrosis, malignant bone marrow infiltration, solid tumors, and/or patellofemoral dysplasia based on clinical assessment, or imaging
* Known autoimmune disease with inflammatory arthritis (including but not limited to rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus), crystal-induced arthritides (gout or pseudogout arthritis), active acute or chronic infection of the knee joint, Lyme disease involving the knee, reactive arthritis, systemic cartilage disorders, moderate to severe fibromyalgia, a known systemic connective tissue disease or a widespread pain index >4.
* Inability to undergo MRI (e.g., claustrophobia, body size, leg not fitting in the coil) or contraindications to MRI (e.g., non MRI-compatible metallic implants, metallic foreign bodies, pacemaker, defibrillator)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cartilage volume in the index region of the target knee by magnetic resonance imaging at Week 52 | Baseline and Week 52
  Change in cartilage volume in certain regions in the knee measured by magnetic resonance imaging at Week 52 compared to the volume prior to receiving RHH646
Number of participants with Adverse Events | From start of treatment until study completion (approximately 14 months)
  Adverse events and clinically notable findings in vital signs, ECG, hematology, blood chemistry, and urinalysis

SECONDARY OUTCOMES:
RHH646 plasma concentrations | Baseline, up to End of Study visit (approximately month 13)
  Concentration of RHH646 in plasma

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Clinical Trials Research, Lincoln, California
  - Conquest Research, Winter Park, Florida
  - Clinical Trial Network, Houston, Texas
  - Pioneer Research Solutions, Sugar Land, Texas
- Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires, Argentina
- Denmark (2):
  - Novartis Investigative Site, Gandrup
  - Novartis Investigative Site, Herlev
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Santiago de Compostela, A Coruna, Spain

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com